CLINICAL TRIAL: NCT07402200
Title: Disrupting Noxious Synergies of Indoor Air Pollutants and Their Impact in Childhood Health and Wellbeing, Using Advanced Intelligent Multisensing and Green Interventions: an Interventional Study in a Sub-group of Schoolchildren
Brief Title: Study of Indoor Air Pollutants and Their Impact in Children's Health and Wellbeing
Acronym: SynAir-G2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL23_0262; 2024-A00254-43 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2026-01-19; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Allergy
Keywords: Air pollution; asthma; allergy
MeSH Terms: conditions — Hypersensitivity; Asthma | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Other): Subjects who have previously declared to suffer from asthma and/or allergic rhinitis and/or other allergic diseases (cases)
  Interventions: Other: Standardized questionnaires; Other: Lung function tests; Diagnostic Test: Prick tests; Other: Biological samples; Device: Portable sensors
- Control group (Other): Subjects who have previously declared not presenting any allergic/respiratory symptoms (healthy controls)
  Interventions: Other: Standardized questionnaires; Other: Lung function tests; Diagnostic Test: Prick tests; Other: Biological samples; Device: Portable sensors

INTERVENTIONS:
Other: Standardized questionnaires — Baseline questionnaires for cases and follow-up questionnaires for cases and controls will be completed to collect data on sociodemographic characteristics, health outcomes, potential risk factors, lifestyle, and living environment.
Other: Lung function tests — All participants, including cases and controls, will undergo comprehensive spirometry testing, pulse oximetry assessment, and fractional exhaled nitric oxide (FeNO) measurement.
Diagnostic Test: Prick tests — Cases and controls will undergo skin prick testing for common allergens, including house dust mites, cat, dog, Alternaria, cypress, birch, plane tree (Platanus), grass, latex, olive tree, ragweed, and mugwort,...
Other: Biological samples — Subjects and their parents/guardians will be given the option to provide blood, urine, and nasopharyngeal samples.
Device: Portable sensors — Up to 10 subjects ( with their parents/guardians consent) will be given the option to use CANARIN devices, to monitor at the individual level exposures to air pollutants (PM and VOC) and other environmental factors (temperature, humidity, pressure) in and outside school.

SUMMARY:
The goal of this study is to identify and assess in real time the impact of the combined action of various types of air and dust pollutants within a classroom on children's health and quality of life, particularly regarding atopic/allergic diseases in children, and on potential exposure to pollutants at home.

Participants will answer questionnaires regarding their health and medications, undergo allergy tests, perform non-invasive lung function tests and check blood oxygen levels.

DETAILED DESCRIPTION:
The number and types of indoor air pollutants in schools is rising, however little is known about the impact of their potentially synergistic interactions, upon schoolchildren health. Among children, highly susceptible individuals to air pollution include allergy and asthma sufferers, and a low socioeconomic background, however no specific guidance is available.

The design of the study provides a unique setting to prospectively assess the synergistic effect of pollutants at school and outdoor on several health aspects in a large and diverse cohort. Most importantly, the continuous nature of information provided by sentinel devices will provide an individualized baseline of specific indicators that will be monitored during the follow up period, to identify personalized health alterations, instead of comparing to generalized standards. Health outcome data, including respiratory health, immune fitness and both mental and non-mental perspectives, focusing on asthmatic/allergic children, will contribute to pollution sensing in an iterative way

ELIGIBILITY:
Inclusion Criteria:

* Child included in the SynAir-G observational study
* Child and caregiver(s) willing to follow the study procedures
* Written informed consent from the child's parents/guardians
* For case group, at least one positive answer (yes) to any of the following questions and for control group, negative answers to all the following questions based on the baseline questionnaire administered in the SynAir-G observational study, as shown below.:

  a. General health i. Does your child have any health problems (if yes to asthma, allergic rhinitis /rhino-conjunctivitis, atopic dermatitis)? b. Asthma i. Has your child ever had wheezing or whistling in the chest in the past 12 months? ii. In the past 12 months, has your child's chest sounded wheezy during or after exercise? iii. In the past 12 months, has your child had a dry cough at night, apart from a cough associated with a cold or chest infection? c. Rhinitis i. In the past 12 months has your child had a problem with sneezing, or a runny, or blocked nose when she/he DID NOT have a cold or the flu? d. Eczema (both answers yes) i. Has your child had this itchy rash at any time in the past 12 months? If so, has this itchy rash at any time affected any of the following places: the folds of the elbows, behind the knees, in front of the ankles, under the buttocks, or around the neck, ears or eyes? e. Food allergy i. Has your child had diagnosed food allergy during last 12 months?
* For case group: Diagnosis of asthma/allergic rhinitis/eczema/food allergy (based on SYNAIR-G baseline questionnaire), active during the past year.
* For control group: absence of diagnosis of asthma/allergic rhinitis/eczema/food allergy (based on SYNAIR-G baseline questionnaire)

Exclusion Criteria:

* Child or child's parents/guardians who:

  1. Refuse to participate in the project / to give informed consent.
  2. Do not want to follow the protocol procedures.
  3. Do not read or/and write in French.
  4. Plan a long stay outside the region that does not allow them to follow the visit plan.
  5. The child is not affiliated to the French social security service

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Statistically significant differences in spirometric parameter, Peak Flow, between case and control groups | 10 Months
  Assessment of peak expiratory flow (Peak Flow, defined as the maximum flow achieved during a forced expiration, measured in L/min) between cases and controls in relation to air and dust contaminants, as assessed in the SynAirG observational study
Statistically significant differences in FeNO measurements between case and control groups | 10 Months
  Evaluation of statistically significant differences in fractional exhaled nitric oxide (FeNO, the concentration of nitric oxide in exhaled breath, measured in parts per billion [ppb]) between cases and controls in relation to air and dust contaminants, as assessed in the SynAirG observational study
Evaluation of statistically significant differences in spirometric parameter, FEV, between case and control groups | 10 months
  Assessment of Forced expiratory volume in 1 second (FEV₁, defined as the volume exhaled during the first second of a forced expiration, measured in L) comparing case and control groups with respect to air and dust contaminants, as assessed in the SynAirG observational study
Evaluation of statistically significant differences in spirometric parameter, FVC, between case and control groups | 10 months
  Assessment of forced vital capacity (FVC, defined as the total volume forcibly exhaled after full inspiration, measured in L), comparing case and control groups with respect to air and dust contaminants within the SynAirG observational study
Statistically significant differences in the spirometric parameter, FEV₁/FVC ratio, between case and control groups | 10 months
  Assessment of the FEV₁/FVC ratio (the proportion of FVC exhaled in the first second, measured in %), between cases and controls in relation to air and dust contaminants, as assessed in the SynAirG observational study
Statistically significant differences in spirometric parameter, FEF, between case and control groups | 10 months
  Assessment of forced expiratory flow at 25%, 50%, and 75% of FVC (FEF₂₅, FEF₅₀, and FEF₇₅, instantaneous expiratory flow rates at the corresponding lung volumes, measured in L/s), between cases and controls in relation to air and dust contaminants, as assessed in the SynAirG observational study
Evaluation of statistically significant differences in spirometric parameter, mean forced expiratory flow, between case and control groups | 10 months
  Assessment of mean forced expiratory flow between 25% and 75% of FVC (FEF₂₅-₇₅, the average expiratory flow over the middle portion of forced expiration, measured in L/s), between cases and controls in relation to air and dust contaminants, as assessed in the SynAirG observational study

SECONDARY OUTCOMES:
Disease control in asthma and allergies in relation to air and dust contaminants | 10 Months
  Evaluation of statistically significant differences in disease control (for asthma and allergic rhinitis and other allergies) between cases, in relation to air and dust contaminants as assessed in the SynAirG observational study
Statistically significant differences in biological biomarkers between case and control groups | 10 Months
  Evaluation of statistically significant differences in biological biomarkers (blood, urine, nasopharyngeal samples) between cases and controls, in relation to air and dust contaminants as assessed in the SynAirG observational study

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France